CLINICAL TRIAL: NCT00192764
Title: Phase II Study of Short High-dose CHOP Chemotherapy for Aggressive Non-Hodgkin's Lymphoma
Brief Title: High Dose CHOP in Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RonHDCHOP.CTIL
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: large cell lymphoma; CHOP; cyclophosphamide; high-dose
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Dendritic Cell Sarcoma, Interdigitating | interventions — Cyclophosphamide

INTERVENTIONS:
Drug: high-dose cyclophosphamide

SUMMARY:
The study hypothesis is that intensification of CHOP by dose escalation of the most active drugs in the combination will improve treatment outcome. Patients with diffuse large-cell lymphoma are treated by high cyclophosphamide containing CHOP. The planned dose is 3000 mg/m2 which is 4 times the atandard one. Only 4 cycles are given.

ELIGIBILITY:
Inclusion Criteria:

* large-cell non-Hodgkin's lymphoma
* IPI low-intermediate, high-intermediate and high or bulky mediastinum
* age 18-65

Exclusion Criteria:

* previous treatment for lymphoma
* serious concurrent systemic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 1996-12; Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Failure-free survival

SECONDARY OUTCOMES:
overall survival
response rate
toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ron Epelbaum, MD, Principal Investigator — nonaffiliated
Locations (1):
- Department of Oncology, Rambam Medical Center, Haifa, Israel